CLINICAL TRIAL: NCT02778945
Title: Deep Versus Moderate Neuromuscular Blockade for Optimising Surgical Conditions Include Patient Benefits During Spinal Surgery: A Randomized Controlled Double Blinded Clinical Study
Brief Title: Neuromuscular Blockade for Optimising Surgical Conditions During Spinal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Chon Jin Young, Professor, Department of Anesthesiology and Pain Medicine, The Catholic University of Korea, College of Medicine,, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ANESTHA-NMB1
Record Dates: First submitted 2016-04-22; First posted 2016-05-20 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Neuromuscular Block; Orthopedic Disorder of Spine; Muscle Weakness
Keywords: spinal surgery; sugammadex; deep neuromuscular block; shear wave elastography; neuromuscular monitoring
MeSH Terms: conditions — Muscle Weakness | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group D (Deep NMB group) (Experimental): Neuromuscular block with Rocuronium 0.9 mg/kg for anesthetic induction Infusion of Rocuronium 0.3mg/kg/hr titrated to maintain a post-tetanic count (PTC)0-2 during the operation.
  Interventions: Drug: Rocuronium 0.9 mg/kg
- Group I (Intermediate NMB group) (Active Comparator): Use NMB as conventional clinical usage Neuromuscular block with Rocuronium 0.6 mg/kg for anesthetic induction Intermittent bolus i.v injection of Rocuronium 0.15mg/kg for train-of-four (TOF) 1-2 during the operation
  Interventions: Drug: Rocuronium 0.6 mg/kg

INTERVENTIONS:
Drug: Rocuronium 0.9 mg/kg — Neuromuscular block with Rocuronium 0.9 mg/kg for anesthetic induction Infusion of Rocuronium 0.3mg/kg/hr titrated to maintain a post-tetanic count (PTC)0-2 during the operation.
  Arms: Group D (Deep NMB group)
Drug: Rocuronium 0.6 mg/kg — Neuromuscular block with Rocuronium 0.6 mg/kg for anesthetic induction Intermittent bolus i.v injection of Rocuronium 0.15mg/kg for train-of-four (TOF) 1-2 during the operation
  Arms: Group I (Intermediate NMB group)

SUMMARY:
In the present study, the investigators compare intermediate and deep NMB i.e. the two extreme regimes of muscle paralysis (neuromuscular block; NMB), (I) patients receiving intermediate muscle paralysis (''control, conventional NMB'') versus (II) patients with a deep neuromuscular blockade with rocuronium (''Deep NMB''), will be compared during a surgical procedure which is considered to be very sensitive for inadequate muscle relaxation, elective minimally invasive spinal surgery.

The primary objective of this trial is to compare the operation time reduction with the help of the decreased stiffness of targeted back muscle surrounding the surgical field.

The changed back muscle stiffness also measured as secondary objective goal by a mechanical tension weighing scale and also taking ultrasonography using shear wave elastography (SWE).

Other observational objectives are divided into the following categories of stakeholders: patients, surgeons and anesthesiologists', done by collecting the variety of clinical parameters. The following will be collected and compared.

1. For patients Intraoperative radiation amount, post-anesthetic care unit(PACU) stay, transfer rate to SICU for post-op. care, post-operative respiratory complication rate, and total hospital costs.
2. For surgeons Post-operative complications in regard to operation field, and evaluate surgical conditions using a Visual Analogue Scale(VAS score) in surgeon's side.
3. For anesthesiologists Intraoperative ventilation parameters of patients, and evaluate surgical conditions using a Visual Analogue Scale(VAS score) in anesthesiologist's side.

DETAILED DESCRIPTION:
All patients will be randomly assigned to two groups after IRB (institutional review board) approval, receiving either deep neuromuscular blockade (''Deep NMB'') or intermediate neuromuscular block (''Control NMB''). Enrolled patients will be given a number in sequence of their enrollment and received a treatment code using a randomization schedule.

The team taking care of patient perioperatively will be blinded regarding the study; this included the surgeons (This study use two different responsible surgeon attendings) and their team, the anesthesia care team in the operating room, in the PACU and the pain physician responsible for postoperative pain management (same as the protocols of the departmental and hospital clinical process).

An additional unblinded anesthesiologist involved in the study management will present from patients' arrival in the operation room to the patients' discharge from the PACU. The unblinded study anesthesiologist takes care of the patients' anesthesia induction, calibration and documentation of the neuromuscular monitoring and the management of the neuromuscular blockade.

Primary endpoint:

To compare the measurements of the operation time reduction, the operation time should be recorded by institutional electronic medical chart from the incision to the final suture closure of surgical wound. A difference of 10% change of operation time between two groups is considered of clinically meaningful difference.

Secondary endpoints:

By using Mechanical Tension Weighing Scale (MTWS) of mechanical dynamometer and also Shear Wave Ultrasound Elastography(SWE), values are taken as followings.

1. Shear Wave Ultrasound Elastography(SWE):

   SWE score value will be collected 3 times as followings. First, After enrolled, the obtained informed consent for this clinical study and screening, SWE score measure will be taken prior to surgery as a basal value from the patient.

   Second, After Induction and patient positioning, measure the targeted back muscle stiffness by using ultrasonography of SWE.

   Third, SWE score measure finally after the stich out before the discharge.
2. Mechanical Tension Weighing Scale(MTWS) of mechanical dynamometer:

After surgical incision, measure the targeted back muscle stiffness by using MTWS. It will be compared between the study groups.

Other check points:

To compare the safety and benefits of deep neuromuscular block over intermediate conventional NMB with corresponding sugammadex reversal.

(Other check points might be changed before the clinical trial initiation circumstantially)

The other check point variables will be collected for investigating to compare the safety and benefits which are divided into patients, surgeons and anesthesiologists' ones by collecting the variety of clinical parameters.

1. For patients intraoperative radiation amount, operation duration, anesthesia duration, post-anesthetic care unit(PACU) stay, transfer rate to SICU for post-op. care, post-operative respiratory complication rate, post-op pain score include patient controlled analgesia(PCA), post-op nausea and vomiting(PONV), and total hospital costs.
2. For surgeons unintended movements during surgery, compromised operating field by tense surrounding muscles, post-operative complications in regard to operation field, and evaluate surgical conditions using a Visual Analogue Scale(VAS score) which will be correlated with muscle stiffness measure by weighing scale and SWE.
3. For anesthesiologists Anesthetic time, intraoperative ventilation parameters of patients, intraoperative vital sign monitor values, and evaluate surgical conditions using a Visual Analogue Scale(VAS score) which will be correlated with muscle stiffness measure by weighing scale and SWE.

All clinical parameters will be collected within 48 hours after surgery except the total hospital costs of the patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients had to be scheduled by the surgeons for an elective spinal surgery required correction of 1 to 3 segment level of spine under general anesthesia.
* Patients with ASA-classification (the American Society of Anesthesiologists) physical status classed as I to II aged 19 years old and over will be enrolled.

Exclusion Criteria:

* expected a difficult airway
* known neuromuscular disease
* known allergy or hypersensitivity to one of the drugs used in this study
* intake of any medication that might interact with muscle relaxants.
* Female subjects will be excluded if they were either pregnant, of childbearing potential, not using a mechanical method of birth control, or if they were breast-feeding.
* subjects who are unable to understand or successfully administer a patient controlled analgesia (PCA) device,
* subjects who are declined to participate during the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
the operation time | Intraoperative
  Primary endpoint:
  To compare the measurements of the operation time reduction, the operation time should be recorded by institutional electronic medical chart from the incision to the final suture closure of surgical wound. A difference of 10% change of operation time between two groups is considered of clinically meaningful difference.

SECONDARY OUTCOMES:
back muscle stiffness ( 1. Shear Wave Ultrasound Elastography(SWE) ) | Intraoperative
  1. Shear Wave Ultrasound Elastography(SWE): SWE score value will be collected 3 times as followings. First, After enrolled, the obtained informed consent for this clinical study and screening, SWE score measure will be taken prior to surgery as a basal value from the patient.
  Second, After Induction and patient positioning, measure the targeted back muscle stiffness by using ultrasonography of SWE.
  Third, SWE score measure finally after the stich out before the discharge.
back muscle stiffness (2.Mechanical Tension Weighing Scale (MTWS) of mechanical dynamometer) | Intraoperative
  2. Mechanical Tension Weighing Scale(MTWS) of mechanical dynamometer: After surgical incision, measure the targeted back muscle stiffness by using MTWS. It will be compared between the study groups.

OTHER OUTCOMES:
post-anesthetic care unit stay | 1 hour after operation
  time duration during post-anesthetic care unit stay
transfer rate to intensive care unit | 1 hour after operation
post-op pain score | 30minutes, 6hours, 12hours, 48hours after operation
  post operative pain is measured when 30 minutes, 6 hours, 12 hours, 24 hours, 48 hours postoperatively using visual analogue scale.
post-op nausea and vomiting(PONV) | 30minutes, 6hours, 12hours, 48hours after operation
  post operative nausea and vomiting is measured when 30 minutes, 6 hours, 12 hours, 24 hours, 48 hours postoperatively using visual analogue scale.
total hospital cost | 4 weeks after operation
  calculated in KRW
surgical condition | Intraoperative
  evaluate surgical conditions using a Visual Analogue Scale(VAS score) asked to surgeon and anesthesiologist, respectively.
intraoperative ventilation parameters (1. lung compliance) | Intraoperative
  lung compliance is measured by anesthetic machine ( GE Avance)
intraoperative ventilation parameters (2. peak airway pressure) | Intraoperative
  peak pressure is measured by anesthetic machine ( GE Avance)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Young Chon, M.D., Ph.D., Study Chair — Department of Anesthesiology and pain medicine, Yeouido St. Mary's Hospital
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fryer G, Morris T, Gibbons P. Paraspinal muscles and intervertebral dysfunction: part two. J Manipulative Physiol Ther. 2004 Jun;27(5):348-57. doi: 10.1016/j.jmpt.2004.04.008. PMID 15195042
- [Background] Brouwer PA, Brand R, van den Akker-van Marle ME, Jacobs WC, Schenk B, van den Berg-Huijsmans AA, Koes BW, van Buchem MA, Arts MP, Peul WC. Percutaneous laser disc decompression versus conventional microdiscectomy in sciatica: a randomized controlled trial. Spine J. 2015 May 1;15(5):857-65. doi: 10.1016/j.spinee.2015.01.020. Epub 2015 Jan 20. PMID 25614151
- [Background] Li YL, Liu YL, Xu CM, Lv XH, Wan ZH. The effects of neuromuscular blockade on operating conditions during general anesthesia for spinal surgery. J Neurosurg Anesthesiol. 2014 Jan;26(1):45-9. doi: 10.1097/ANA.0b013e31829f3805. PMID 23887680
- [Background] Carron M. Respiratory benefits of deep neuromuscular block during laparoscopic surgery in a patient with end-stage lung disease. Br J Anaesth. 2015 Jan;114(1):158-9. doi: 10.1093/bja/aeu419. No abstract available. PMID 25500396
- [Background] Eichel L, Batzold P, Erturk E. Operator experience and adequate anesthesia improve treatment outcome with third-generation lithotripters. J Endourol. 2001 Sep;15(7):671-3. doi: 10.1089/08927790152596217. PMID 11697394
- [Background] Mergeay M, Verster A, Van Aken D, Vercauteren M. Regional versus general anesthesia for spine surgery. A comprehensive review. Acta Anaesthesiol Belg. 2015;66(1):1-9. PMID 26103736
- [Background] Simons GD, Mense S. Understanding and measurement of muscle tone as related to clinical muscle pain. Pain. 1998 Mar;75(1):1-17. doi: 10.1016/S0304-3959(97)00102-4. PMID 9539669
- [Background] Buchmann J, Neustadt B, Buchmann-Barthel K, Rudolph S, Klauer T, Reis O, Smolenski U, Buchmann H, Wagner KF, Haessler F. Objective measurement of tissue tension in myofascial trigger point areas before and during the administration of anesthesia with complete blocking of neuromuscular transmission. Clin J Pain. 2014 Mar;30(3):191-8. doi: 10.1097/AJP.0b013e3182971866. PMID 23689350
- [Background] de Paula Simola RA, Harms N, Raeder C, Kellmann M, Meyer T, Pfeiffer M, Ferrauti A. Assessment of neuromuscular function after different strength training protocols using tensiomyography. J Strength Cond Res. 2015 May;29(5):1339-48. doi: 10.1519/JSC.0000000000000768. PMID 25474337
- [Background] van Ramshorst GH, Salih M, Hop WC, van Waes OJ, Kleinrensink GJ, Goossens RH, Lange JF. Noninvasive assessment of intra-abdominal pressure by measurement of abdominal wall tension. J Surg Res. 2011 Nov;171(1):240-4. doi: 10.1016/j.jss.2010.02.007. Epub 2010 Mar 5. PMID 20462598
- [Background] Oliva-Pascual-Vaca A, Heredia-Rizo AM, Barbosa-Romero A, Oliva-Pascual-Vaca J, Rodriguez-Blanco C, Tejero-Garcia S. Assessment of paraspinal muscle hardness in subjects with a mild single scoliosis curve: a preliminary myotonometer study. J Manipulative Physiol Ther. 2014 Jun;37(5):326-33. doi: 10.1016/j.jmpt.2014.03.001. PMID 24928641
- [Background] Hamzat TK. Physical characteristics as predictors of quadriceps muscle isometric strength: a pilot study. Afr J Med Med Sci. 2001 Sep;30(3):179-81. PMID 14510124
- [Background] Bercoff J, Tanter M, Fink M. Supersonic shear imaging: a new technique for soft tissue elasticity mapping. IEEE Trans Ultrason Ferroelectr Freq Control. 2004 Apr;51(4):396-409. doi: 10.1109/tuffc.2004.1295425. PMID 15139541
- [Background] Brandenburg JE, Eby SF, Song P, Zhao H, Landry BW, Kingsley-Berg S, Bamlet WR, Chen S, Sieck GC, An KN. Feasibility and reliability of quantifying passive muscle stiffness in young children by using shear wave ultrasound elastography. J Ultrasound Med. 2015 Apr;34(4):663-70. doi: 10.7863/ultra.34.4.663. PMID 25792582
- [Background] Lacourpaille L, Hug F, Guevel A, Pereon Y, Magot A, Hogrel JY, Nordez A. Non-invasive assessment of muscle stiffness in patients with Duchenne muscular dystrophy. Muscle Nerve. 2015 Feb;51(2):284-6. doi: 10.1002/mus.24445. Epub 2014 Dec 23. PMID 25187068
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Baykara N, Sahin T, Alpar R, Solak M, Toker K. Evaluation of intense neuromuscular blockade caused by rocuronium using posttetanic count in male and female patients. J Clin Anesth. 2003 Sep;15(6):446-50. doi: 10.1016/s0952-8180(03)00110-7. PMID 14652123
- [Background] Takagi S, Ozaki M, Iwasaki H, Hatano Y, Takeda J. [Effects of sevoflurane and propofol on neuromuscular blocking action of Org 9426 (rocuronium bromide) infused continuously in Japanese patients]. Masui. 2006 Aug;55(8):963-70. Japanese. PMID 16910475